CLINICAL TRIAL: NCT03059446
Title: Open-label Rollover Study of Cenicriviroc for the Treatment of Liver Fibrosis in Adult Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Rollover Study of Cenicriviroc for the Treatment of Liver Fibrosis in Participants With Nonalcoholic Steatohepatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to lack of efficacy based on the results of Part I of the AURORA study.
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3152-201-002; 2016-004754-15 (EudraCT Number)
Record Dates: First submitted 2017-02-03; First posted 2017-02-23 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-09

CONDITIONS: Nonalcoholic Steatohepatitis; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — cenicriviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cenicriviroc (CVC) 150 mg (Experimental): Cenicriviroc 150 mg tablet once daily in the morning with food until the study was terminated (up to approximately 4 years).
  Interventions: Drug: Cenicriviroc

INTERVENTIONS:
Drug: Cenicriviroc — Cenicriviroc immediate release tablets
  Other Names: CVC

SUMMARY:
This rollover study will provide open-label treatment with cenicriviroc and will assess the long-term safety of continued treatment with cenicriviroc in participants who participated in either the CENTAUR study 652-2-203 [NCT02217475] or the AURORA study [NCT03028740].

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of both Treatment Period 1 and Treatment Period 2, of the CENTAUR Study (652-2-203), including a Year 2 liver biopsy.
* Completed the AURORA study (3152-301-002) as a result of reaching an adjudicated liver-related clinical outcome in Part 1 or Part 2 of the study of:
* Histopathological progression to cirrhosis
* Model for end-stage liver disease (MELD) score ≥ 15
* Ascites (requiring intervention, ie, large volume paracentesis ≥ 1L or initiation of a diuretic)
* Hospitalization (as defined by a stay of ≥ 24 hours) for onset of variceal bleed, hepatic encephalopathy (defined by a West Haven Stage of ≥ 2), spontaneous bacterial peritonitis (confirmed by diagnostic paracentesis with positive ascitic fluid bacterial culture).

Exclusion Criteria:

* Prior or planned liver transplantation
* Other know causes of chronic liver disease such as: Alcoholic liver disease, Primary biliary cirrhosis, Primary sclerosing cholangitis, Autoimmune hepatitis, Wilson's disease, hemochromatosis, or iron overload, or Alpha-1 antitrypsin (A1AT) deficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo B Martins, Study Director — Allergan
Locations (71):
- United States (41):
  - Digestive Health Specialists of the Southeast - Dothan, Dothan, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Franco Felizarta, MDv, Bakersfield, California
  - University of California, San Diego (UCSD), La Jolla, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California, San Diego (UCSD) - Medical Center, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Upland Clinical Research, Upland, California
  - Island View Gastroenterology Associates, Ventura, California
  - University of Miami - Schiff Center for Liver Diseases, Miami, Florida
  - Advanced Medical Research, Port Orange, Florida
  - Florida Health Sciences Center, Inc. d/b/a Tampa General Hospital, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Kansas Medical Clinic PA, Topeka, Kansas
  - Delta Research Partners, Llc, Bastrop, Louisiana
  - Tandem Clinical Research LLC, Marrero, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - Mercy Medical Center - Baltimore, Maryland, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Digestive Health Specialists, Tupelo, Mississippi
  - University of Buffalo - Erie County Medical Center, Buffalo, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Wake Research Associates, LLC - Raleigh, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Consultants for Clinical Research - Cincinnati, Cincinnati, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - ClinSearch LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Digestive Health Research, Lebanon, Tennessee
  - The University of Texas - Health Science Center & Medical School at Houston, Houston, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University Medical College of Virginia, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (5):
  - Royal Brisbane Hospital and Women's Hospital, Herston, Queensland
  - Central Adelaide Local Health Network Inc - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
- Belgium (3):
  - University Hospital Erasmus (Brussels), Brussels
  - UCL Saint Luc Bruxelles, Brussels
  - Antwerp University Hospital (UZA), Edegem
- France (3):
  - CHU Angers, Angers
  - Hopital Saint Antoine, Paris
  - Purpan CHU Toulouse, Toulouse
- Germany (7):
  - Uniklinik RWTH Aachen, Aachen
  - Charite - University Hospital Berlin - Campus Virchow - Hospital, Berlin
  - Uniklinik Koeln, Poliklinik fuer Endokrinologie, Diabetologie und Praeventivmedizin (ZEDP), Cologne
  - Universitaetsklinikum Hamburg-Eppendorf - I. Medizinische Klinik und Poliklinik, Hamburg
  - Universitaetsklinikum Heidelberg - Innere Medizin IV, Heidelberg
  - Eugastro GmbH, Leipzig
  - University Hospital Giessen and Marburg GmbH, Marburg
- Prince of Wales Hospital, Shatin, Hong Kong
- Italy (3):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - AOU Policlinico Paolo Giaccone di Palermo, Palermo
- Poland (2):
  - ID Clinic, Mysłowice
  - Centrum Badan Klinicznych Piotr Napora Lekarze Sp. p., Wroclaw
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
- United Kingdom (2):
  - Nottingham NHS Treatment Centre, Nottingham
  - Queen Alexandra Hospital, Portsmouth

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the CENTAUR study [NCT02217475] or the AURORA study [NCT03028740] were eligible for enrollment in this rollover study.
Period: Overall Study
Arm/Group | Cenicriviroc (CVC) 150 mg
Started | 167
Completed | 0
Not Completed | 167
Not completed — Adverse Event | 11
Not completed — Withdrawal of Consent | 16
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 1
Not completed — Study Terminated by Sponsor | 131
Not completed — Reason not Specified | 5

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of study drug.
Arm/Group | Cenicriviroc (CVC) 150 mg
Number analyzed (Participants) | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 143
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 4
  White | 150
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. A treatment-emergent AE is an AE that occurs after a participant receives study drug.
Time Frame: Day 1 until the study was terminated (up to approximately 4 years)
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenicriviroc (CVC) 150 mg
Number analyzed (Participants) | 167
Participants | 140

ADVERSE EVENTS:
Time Frame: Day 1 until the study was terminated (Up to approximately 4 years)
Arm/Group | Cenicriviroc (CVC) 150 mg
All-Cause Mortality (participants affected / at risk) | 1/167
Serious Adverse Events (participants affected / at risk) | 40/167
Other Adverse Events (participants affected / at risk) | 98/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cenicriviroc (CVC) 150 mg (N=167)
Angina pectoris (Cardiac disorders) | 3
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Salivary gland calculus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 3
Pneumonia legionella (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Bone abscess (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Carbuncle (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Q fever (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Post procedural fever (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Gout (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/88 — Number of participants at risk is based on the female population.
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Migraine with aura (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Uraemic encephalopathy (Nervous system disorders) | 1
Vertebral artery stenosis (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphatic fistula (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cenicriviroc (CVC) 150 mg (N=167)
Diarrhoea (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 10
Nasopharyngitis (Infections and infestations) | 17
Influenza (Infections and infestations) | 14
Bronchitis (Infections and infestations) | 12
Sinusitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 9
Alanine aminotransferase increased (Investigations) | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-04-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT03059446/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT03059446/SAP_001.pdf